CLINICAL TRIAL: NCT02051868
Title: An International Multicentre Open Label Randomised Phase II Advanced Anal Cancer Trial Comparing Cisplatin Plus 5 FU vs Carboplatin Plus Weekly Paclitaxel in Patients With Inoperable Locally Recurrent or Metastatic Disease
Brief Title: International Multicentre Study in Advanced Anal Cancer Comparing Cisplatin Plus 5 FU vs Carboplatin Plus Weekly Paclitaxel
Acronym: InterAACT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); Australasian Gastro-Intestinal Trials Group (Network); ECOG-ACRIN Cancer Research Group (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network); International Rare Cancers Initiative (IRCI ) This study is indorsed by IRCI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR 3847 InterAACT; 2013-001949-13 (EudraCT Number)
Record Dates: First submitted 2014-01-13; First posted 2014-01-31 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Squamous Cell Carcinoma of the Anus
Keywords: Squamous cell carcinoma of the anus; Anal cancer; Cancer of the anus; SCCA; Cisplatin-5FU; Carboplatin-Paclitaxel; inoperable; locally recurrent; metastatic
MeSH Terms: conditions — Anus Neoplasms; Neoplasm Metastasis | interventions — Cisplatin; Fluorouracil; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Cisplatin and 5-Fluorouracil
  Interventions: Drug: Cisplatin; Drug: 5-Fluorouracil (5-FU)
- Arm B (Experimental): Carboplatin plus Paclitaxel
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 60 mg/m2 as a 1 hour i.v. infusion once every 3 weeks.
  Other Names: Systematic (IUPAC) name: (SP-4-2)-diamminedichloridoplatinum; CAS number 15663-27-1 Y; ATC code L01XA01
  Arms: Arm A
Drug: 5-Fluorouracil (5-FU) — 5-FU 1000 mg/m2/24h as a 96-hour continuous infusion over days 1 to 4 every 3 weeks.
  Other Names: Systematic (IUPAC) name: 5-fluoro-1H,3H-pyrimidine-2,4-dione; CAS number 51-21-8 Y; ATC code L01BC02
  Arms: Arm A
Drug: Carboplatin — Carboplatin 1-hour i.v. infusion to an area under the curve (AUC) of 5 once every 4 weeks.
  Other Names: Systematic (IUPAC) name: cis-diammine(cyclobutane-1,1-dicarboxylate-O,O')platinum(II); CAS number 41575-94-4 Y; ATC code L01XA02
  Arms: Arm B
Drug: Paclitaxel — Paclitaxel 80 mg/m2 as a 1-hour i.v. infusion on day 1,8 and 15 of each (4-weekly) cycle.
  Other Names: (2α,4α,5β,7β,10β,13α)-4,10-bis(acetyloxy)-13-{[(2R,3S)- 3-(benzoylamino)-2-hydroxy-3-phenylpropanoyl]oxy}- 1,7-dihydroxy-9-oxo-5,20-epoxytax-11-en-2-yl benzoate; CAS number 33069-62-4 Y; ATC code L01CD01
  Arms: Arm B

SUMMARY:
Anal cancer is a relatively uncommon disease and there is currently no standard chemotherapy treatment for patients with inoperable locally recurrent or metastatic disease. The aim of this phase II study is compare two well known and largely used chemotherapy regimens - Cisplatin plus 5-fluorouracil vs Carboplatin plus Paclitaxel. The result of this study will set a standard of care for this disease and provide useful information for future Phase III trials.

DETAILED DESCRIPTION:
Study design: This is an international, multicentre, open label, randomised phase II trial. Patients will be randomised to receive either cisplatin plus 5-FU or carboplatin plus weekly paclitaxel. Region (Europe, North America, South America & Australia), (Eastern Cooperative Oncology Group- ECOG) ECOG performance status (PS) (0-1 vs. 2), HIV status (positive vs. negative) and extent of disease (locally recurrent vs. metastatic) will be used as stratification factors. Overall response rate is the primary endpoint.

Indication: First line treatment of patients with inoperable locally recurrent or metastatic squamous cell carcinoma of the anus.

Length of study: Recruitment should be completed within 3 years. The estimated recruitment rate is between 4-6 patients per month once it is established at multiple centres.

Primary Objective: To evaluate best overall response rate by 24 weeks post treatment in the cisplatin plus 5-fluorouracil arm versus the carboplatin plus weekly paclitaxel arm

Secondary Objectives: To evaluate: - Progression-free survival - Overall survival - Disease control rate (stable disease or better) at 12 and 24 weeks - Best overall response of metastatic lesions - Toxicity (graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 4) - Quality of Life (using EORTC QLQ-C30 version 3 and EQ-5D-5L questionnaires).

To assess: The feasibility of conducting a multicentre international study on squamous cell carcinoma of the anus and recruit within a reasonable time frame.

Exploratory Objective: Explorative biomarker analysis including the collection of archived tumour tissue and blood sample at baseline and upon progression.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically verified, uni-dimensionally measurable, inoperable, locally recurrent or metastatic squamous cell carcinoma of the anus.
2. Age ≥18 years.
3. ECOG Performance status ≤2.
4. Measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1.
5. Previous definitive chemoradiotherapy is permitted for early stage squamous cell carcinoma of the anus.
6. HIV+ patients will be considered eligible with a CD4 count of ≥200.
7. Adequate cardiac and respiratory function; absolute neutrophil count (ANC) ≥1.5x10^9/l; white blood cell (WBC) count ≥3x10^9/l; platelets >100x10^9/l; haemoglobin (Hb) ≥9g/dl; creatinine clearance >50ml/minute; serum bilirubin ≤1.5x upper limit of normal (ULN); alanine transaminase (ALT)/aspartate transaminase (AST) ≤2.5x ULN; alkaline phosphatase (ALP) ≤3x ULN.
8. Fertile men and women must agree to take adequate contraceptive precautions during, and for at least six months after therapy.
9. Life expectancy of at least 3 months.

Exclusion Criteria

1. Tumours of adenocarcinoma, melanoma, small cell and basal cell histology are excluded.
2. Previous chemotherapy, radiotherapy or other investigational drug for surgically unresectable locally recurrent or advanced squamous cell carcinoma of the anus
3. Current or recent (within 30 days of first study dosing) treatment with another investigational drug or participation in another investigational study.
4. Documented or symptomatic brain metastases and/or central nervous system metastases or leptomeningeal disease.
5. Surgery or palliative radiotherapy within 28 days of randomisation.
6. Clinically significant (i.e. active) cardiac disease (e.g. symptomatic coronary artery disease, uncontrolled cardiac arrhythmia, or myocardial infarction within the last 6 months). Any history of clinically significant cardiac failure.
7. History of interstitial lung disease (e.g. pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan.
8. Lack of physical integrity of the gastro-intestinal tract, malabsorption syndrome (naso-gastric or jejunostomy feeding tube is permitted).
9. Acute hepatitis C and/or chronic active hepatitis B infection.
10. Serious active infection requiring i.v. antibiotics at enrolment.
11. Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
12. Other clinically significant disease or co-morbidity that may adversely affect the safe delivery of treatment within this trial.
13. Known hypersensitivity to any of the study drugs or excipients.
14. Known peripheral neuropathy ≥ grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible).
15. Pre-existing hearing impairment.
16. Patients planning for a live vaccine.
17. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-08 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Best overall response rate by 24 weeks post treatment | 24 weeks
  Best overall response rate is defined as the percentage of patients achieving confirmed partial or complete responses as per RECIST v1.1 by 24 weeks post treatment start in the intention to treat population. Sensitivity analyse will also be performed.

SECONDARY OUTCOMES:
Feasibility of conducting a multicentre, international study on squamous cell carcinoma of the anus and recruiting within a reasonable time frame. | 3 years
  The study will be conducted in approximately 50 international centres. This secondary endpoint will be measured by (i) the proportion of centres that successfully recruit at least one patient and (ii) overall recruitment rate. We anticipate and would be able to confirm feasibility if 80% of the centres fully engaged with the study. The aim would be to recruit 80 patients in 36 months (10 by month 6, 20 by month 12, 50 by month 24 and 80 by month 36).
Toxicity | Toxicity will be analysed once all patients have been followed up for at least 4 weeks post treatment.
  Toxicity will be graded according to the NCI CTCAE Version 4.0
Progression-free survival | PFS will be analysed once all patients have been followed up for at least 12 months post treatment.
  This is calculated from the date of randomisation to the date of confirmed clinical/radiological progression or death from any cause. Patients who are lost to follow-up, withdraw from follow-up or alive and progression free will be censored at the date of last follow-up.
Overall survival | Overall survival will be analysed once all patients have been followed up for at least 12 months post treatment.
  This is calculated from the date of randomisation to the date of death from any cause. Patients, in whom no death is recorded, will be censored at the date they were last seen alive.
Disease control rate | 12 and 24 weeks post treatment start
  Disease control rate is defined as complete response, partial response or stable disease, and will be assessed in accordance with the RECIST criteria v1.1.
Best overall response rate of non-irradiated lesions | 24 weeks post treatment start
  Best overall response of non-irradiated lesions is defined as the percentage of patients achieving confirmed partial response or complete response as per RECIST v1.1 of non-irradiated sites of disease.
Anti-tumour activity and magnitude of tumour response | 24 weeks
  Anti-tumour activity and magnitude of response will be captured by waterfall plot analyses and indicate the percentage change in tumour size from baseline to the time of best response.
Quality of Life | 3 years
  Quality of Life will be evaluated using the EORTC QLQ C30 and EQ-5D-5L questionnaires. The functional and symptomatic scales and global health status from the QLQ C30 and EQ-5D-5L questionnaire will be calculated as per EORTC and EuroQol guidelines, respectively.
Identification of potential tumour biomarker | 3 years
  Archived tumour tissue (if available) and blood sample will be taken at baseline with a repeat blood sample taken upon progression. Patient can enrol in an optional biomarker study where an additional tumour biopsy would be requested when they progress. The aim of this exploratory analysis is to evaluate the expression of tumour biomarkers in the study population and investigate the association of these with treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sheela Rao, MD, FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (3):
- Laura Gagnon, Boston, Massachusetts, United States
- Margot Gorzeman, Sydney, New South Wales, Australia
- Royal Marsden NHS Foundation Trust, London & Sutton, Sutton, United Kingdom

REFERENCES:
- [Derived] Rao S, Sclafani F, Eng C, Adams RA, Guren MG, Sebag-Montefiore D, Benson A, Bryant A, Peckitt C, Segelov E, Roy A, Seymour MT, Welch J, Saunders MP, Muirhead R, O'Dwyer P, Bridgewater J, Bhide S, Glynne-Jones R, Arnold D, Cunningham D. International Rare Cancers Initiative Multicenter Randomized Phase II Trial of Cisplatin and Fluorouracil Versus Carboplatin and Paclitaxel in Advanced Anal Cancer: InterAAct. J Clin Oncol. 2020 Aug 1;38(22):2510-2518. doi: 10.1200/JCO.19.03266. Epub 2020 Jun 12. PMID 32530769